CLINICAL TRIAL: NCT04358965
Title: Evaluating Safety and Efficacy of Tranexamic Acid Versus Vaginal Misoprostol in Reducing Intraoperative Blood Loss During Abdominal Myomectomy
Brief Title: Tranexamic Acid Versus Vaginal Misoprostol in Abdominal Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: misoprostol myomectomy
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Myomectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intravenous tranexamic acid (Experimental): patients were given a single bolus IV injection of 15 mg/kg of TXA 20 minutes before surgical incision plus one vaginal placebo tablet 1 hour before skin incision
  Interventions: Drug: intravenous tranexamic acid
- vaginal misoprostol (Active Comparator): patients will be given one vaginal misoprostol tablet (200 mcg) 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Interventions: Drug: vaginal misoprostol
- placebo (Placebo Comparator): patients will be given one vaginal placebo tablet 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: intravenous tranexamic acid — patients will be given a single bolus IV injection of 15 mg/kg of tranexamic acid (TXA) 20 minutes before surgical incision plus one vaginal placebo tablet 60 minutes before skin incision.
  Arms: intravenous tranexamic acid
Drug: vaginal misoprostol — patients will be given one vaginal misoprostol tablet (200 mcg) 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Arms: vaginal misoprostol
Drug: placebo — patients will be given one vaginal placebo tablet 60 minutes before skin incision and a normal saline IV bolus 20 minutes before surgical incision
  Arms: placebo

SUMMARY:
the aim of the present study is to evaluate safety and efficacy of tranexamic acid versus vaginal misoprostol in reducing intraoperative blood loss during abdominal myomectomy

ELIGIBILITY:
Inclusion Criteria:

* symptomatic fibroids candidate for abdominal myomectomy

Exclusion Criteria:

* myomas candidate for laparoscopic or hysteroscopic myomectomy and allergy or contraindications to misoprostol or tranexamic acid

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2020-10-10 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | one hour
  intraoperative blood loss will be estimated during open myomectomy in mL